CLINICAL TRIAL: NCT02621983
Title: Aerobic Exercise for Cognition in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1897-P; 1I21RX001897-01A1 (NIH); IRB00082701 (Other: IRB)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Exercise; Cognition
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise (Active Comparator): Subjects with a diagnosis of SCZ will complete aerobic exercises consisting of spin classes 3 times a week on a stationary bicycle ergometer. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes by increasing 5 minutes each week for 12 weeks.
  Interventions: Behavioral: Aerobic Exercise
- Balance and Stretching (Active Comparator): Subjects with a diagnosis of SCZ will complete a balance and stretching program consisting of progressive whole body stretching and toning exercises. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes by increasing 5 minutes each week for 12 weeks.
  Interventions: Behavioral: Balance and Stretching

INTERVENTIONS:
Behavioral: Aerobic Exercise — Subjects with a diagnosis of SCZ will complete aerobic exercises consisting of spin classes 3 times a week on a stationary bicycle ergometer. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes by increasing 5 minutes each week for 12 weeks.
  Arms: Aerobic Exercise
Behavioral: Balance and Stretching — Subjects with a diagnosis of SCZ will complete a balance and stretching program consisting of progressive whole body stretching and toning exercises. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes by increasing 5 minutes each week for 12 weeks.
  Arms: Balance and Stretching

SUMMARY:
This study will evaluate the ability of aerobic exercise (AE) to improve cognition in people with schizophrenia. Participants will be randomly assigned to one of two interventions: (1) aerobic exercise class (stationary bicycle, or "spin" class) for up to 45 minutes three times per week for 12 weeks, or (2) balance and stretching class for up to 45 minutes three times per week for 12 weeks.

DETAILED DESCRIPTION:
Schizophrenia (SCZ) is a severe, chronic, and disabling psychotic illness that affects approximately 87,000 Veterans. Previous studies have reported improved short-term memory with AE, but there in a lack of information on cognitive effects of AE in SCZ. The investigators want to determine if twelve weeks of AE training improves cognitive function in Veterans with SCZ.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* maintained on stable doses of outpatient psychiatric medications for at least 30 days
* compliant with outpatient follow-up
* have a stable place to live
* access to transportation to the hospital
* doing less than 20 minutes per week of regular physical activity in the past month

Exclusion Criteria:

* Bipolar disorder;
* active substance dependence within the prior 30 days
* more than 2 psychiatric admissions within the prior six months
* known HIV infection or AIDS
* history of traumatic brain injury
* current seizure disorder
* Alzheimer's disease or other dementia
* clinical history of mild cognitive impairment
* Parkinson's disease
* other current clinically significant neurological disease
* unstable medical condition that would be expected to interfere with fitness training
* significant hearing or visual impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica J. Duncan, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There is a discrepancy between the enrollment number (50) and the participant flow module (38) because 12 participants either failed the initial screening procedures or were unable to be randomized because they didn't complete the baseline visit prior to randomization.
Groups:
- Aerobic Exercise: Subjects with a diagnosis of schizophrenia (SCZ) will complete aerobic exercises consisting of spin classes 3 times a week on a stationary bicycle ergometer. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes by increasing 5 minutes each week for 12 weeks.
  Aerobic Exercise: Subjects with a diagnosis of SCZ will complete aerobic exercises consisting of spin classes 3 times a week on a stationary bicycle ergometer. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes by increasing 5 minutes each week for 12 weeks.
Period: Overall Study
Arm/Group | Aerobic Exercise | Balance and Stretching
Started | 21 | 17
Completed | 9 | 6
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Balance and Stretching | Total
Number analyzed (Participants) | 21 | 17 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 17 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.524 (6.660) | 53.176 (10.273) | 52.816 (8.239)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 16 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 17 | 36
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 17 | 38
400m Walk Time [Mean (Standard Deviation); unit: seconds] — Population: One individual did not complete the 400m walk because of obstacles on the course. Individual then dropped out of the study.
  seconds
    number analyzed (Participants) | 21 | 16 | 37
    (all) | 358.95 (58.022) | 345.38 (57.218) | 353.08 (57.279)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function, Assessed by Scores on the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Cognitive function will be assessed by using the MATRICS Consensus Cognitive Battery (MCCB). It assesses seven key cognitive domains: processing speed, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The MCCB is a battery of tests with a computerized scoring system that produces T-scores, adjusted for age and sex, that are used by the MCCB software to create composite scores. The range of T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better overall cognitive functioning. A higher composite score on the MCCB is indicative of better cognitive function, however there are no clinically significant thresholds. The scores reported below are means +/- standard deviations of these composite scores.
Time Frame: Baseline, 12 weeks
Population: We had significant drop-out during the course of the 12 week exercise paradigm, therefore only 11 from the Aerobic group and 6 from the Balance and Stretching group completed all 12 weeks worth of exercise.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise | Balance and Stretching
Number analyzed (Participants) | 11 | 6
T-score
  Baseline | 24.909 (9.332) | 31.333 (5.989)
  12 Weeks | 27.727 (10.258) | 32.833 (6.113)

2. Secondary Outcome: Change in Functional Ability
Description: Functional ability will be assessed using the University of California San Diego Performance-Based skills assessment (UPSA). The UPSA is a measure of functional ability to perform common activities of daily living. It assess communication, financial, and household skills as well as the ability to manage medication, navigate transportation, and organize and plan an activity. Each measure creates a raw score which is summed to create a composite score. A higher score indicates better functional ability. No clinically significant thresholds. The maximum score an individual could obtain was 87 and the minimum was 0. The score is reported on scale units.
Time Frame: Baseline, 12 weeks
Population: We had many individuals who dropped out during the course of the 12 week exercise program, this leads to the discrepancy in number of participants analyzed when compared to those who were randomized into the two arms of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise | Balance and Stretching
Number analyzed (Participants) | 11 | 6
units on a scale
  Baseline | 58.55 (13.46) | 67.83 (5.42)
  Week 12 | 60.64 (9.89) | 64.16 (9.28)

3. Secondary Outcome: Change in MCCB Scores
Description: Cognitive function will be assessed by using the MATRICS Consensus Cognitive Battery (MCCB). It assesses seven key cognitive domains: processing speed, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The MCCB is a battery of tests with a computerized scoring system that produces T-scores, adjusted for age and sex, that are used by the MCCB software to create composite scores. The range of T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. A higher composite score on the MCCB is indicative of better cognitive function, however there are no clinically significant thresholds. The scores reported below are means +/- standard deviations of these composite scores.
Time Frame: Baseline, 20 weeks
Population: We had significant drop out from baseline measurement to week 20, accounting for the difference in numbers when compared to the total enrolled. We also had two drop out in the Aerobic Exercise group between week 12 and week 20 accounting, which explains the difference in number between the primary outcome and this outcome.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise | Balance and Stretching
Number analyzed (Participants) | 9 | 6
T-score
  Baseline | 24.78 (7.95) | 31.33 (5.99)
  Week 20 | 29.33 (8.12) | 29.5 (7.64)

4. Secondary Outcome: Change in Scores on the University of California San Diego Performance-Based Skills Assessment (UPSA)
Description: as for outcome 2
Time Frame: Baseline, 20 weeks
Population: The numbers will differ from the initial secondary outcome because we had two individuals drop out of the study between the week 12 and week 20 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise | Balance and Stretching
Number analyzed (Participants) | 9 | 6
units on a scale
  Baseline | 57.66 (14.11) | 67.83 (5.42)
  Week 20 | 64.33 (7.60) | 67.33 (8.21)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected while the subject was enrolled in the study, at most a total of 5 months.
Arm/Group | Aerobic Exercise | Balance and Stretching
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/17
Serious Adverse Events (participants affected / at risk) | 3/21 | 1/17
Other Adverse Events (participants affected / at risk) | 2/21 | 2/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise (N=21) | Balance and Stretching (N=17)
Psychiatric Admission (Psychiatric disorders) | 2 (2) | 0 (0)
Hospital Admission (Cardiac disorders) | 0 (0) | 1 (1)
Adverse Medication Reaction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise (N=21) | Balance and Stretching (N=17)
Car Accident (Social circumstances) | 1 (1) | 0 (0)
Claustrophobia (Psychiatric disorders) | 0 (0) | 1 (1)
Muscle fatigue and pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT02621983/Prot_SAP_000.pdf